CLINICAL TRIAL: NCT05470595
Title: A Phase II, Single-arm Trial of Atezolizumab/Platinum/Etoposide for the Treatment of Advanced Large-cell Neuroendocrine Cancer of the Lung
Brief Title: A Single-arm Trial of Atezolizumab/Platinum/Etoposide for the Treatment of Advanced Large-cell Neuroendocrine Cancer of the Lung
Acronym: LCNEC-ALPINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-ALPINE-077; 2024-515902-15-00 (EU CTIS Number); 2020-002683-31 (EudraCT Number)
Record Dates: First submitted 2022-07-13; First posted 2022-07-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Large Cell Neuroendocrine Carcinoma of the Lung
Keywords: Lung Cancer; LCNEC; Neuroendocrine Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Neuroendocrine | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab/Platinum/Etoposide (Experimental): Atezolizumab/Platinum/Etoposide Platinum will be cisplatin or carboplatin at the investigators discretion.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab (IMP) will be added to Platinum/Etoposide (Standard-of-Care). Four cycles of combined immunochemotherapy 3qw will be follows by maintenance with atezolizumab monotherapy until progression.

SUMMARY:
This phase II clinical trial evaluates the efficacy, safety and tolerability of Atezolizumab in addition to standard of care chemotherapy (Platinum/Etoposide) in LCNEC.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Patients with locally advanced or metastatic large-cell neuroendocrine carcinoma of the lung (LCNEC) without curative treatment options (patients with mixed histology are eligible if LCNEC is the predominant histology i.e. ≥50%)
3. Previously untreated with systemic therapy (note: patients relapsing after curative radio chemotherapy or adjuvant chemotherapy are eligible if relapse occurs ≥6 months after discontinuation of curative treatment)
4. Planned treatment with Carboplatin or Cisplatin and Etoposide (SoC)
5. ECOG performance status: 0-2
6. age ≥18 years
7. measurable disease according to RECIST v1.1
8. adequate organ function defined as:

   1. ALAT/ASAT ≤2.5x ULN or ≤3.5x ULN in case of liver metastases
   2. Bilirubin ≤1.5x ULN or ≤2.5x ULN in case of liver metastases
   3. Creatinine ≤1.5x ULN or Creatinine clearance according to Cockroft-Gault >60 ml/min
   4. Neutrophils ≥1 Gpt/l, Platelets >50 Gpt/l unless caused by bone marrow carcinosis

Exclusion Criteria:

1. Symptomatic brain metastases (patients with asymptomatic brain metastases are allowed provided they are stable without steroid treatment for at least 3 weeks)
2. Severe autoimmune disease (patients with endocrine autoimmune disorders are allowed as long as they are on stable substitution treatment)
3. Severe uncontrolled infection
4. Prior treatment with either Atezolizumab or other immune checkpoint inhibitor
5. Any prior treatment for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | appr. 72 months
  To assess the efficacy of Atezolizumab in addition to standard of care chemotherapy (Platinum/Etoposide) in LCNEC as measured by overall survival.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | appr. 72 months
  According to RECIST v1.1 as assessed by local investigator.
Immune Objective Response Rate (iORR) | appr. 72 months
  According to iRECIST as assessed by local investigator.
Disease Control Rate (DCR) | appr. 72 months
  According to RECIST v1.1 as assessed by local investigator.
Progression Free Survival (PFS) | appr. 72 months
Immune Progression Free Survival (iPFS) | appr. 72 months
Duration of Response (DoR) | appr. 72 months
Progression Free Survival (PFS) rate at one year | 1 year
Immune Progression Free Survival (iPFS) rate at one year | 1 year
Overall survival at one year | 1 year
Incidence, intensity, seriousness, relationship to Atezolizumab, and outcome of adverse events graded according to NCI CTCAE (v5.0). | appr. 72 months

OTHER OUTCOMES:
Secondary efficacy endpoints in defined molecular subtypes (NSCLC-type / SCLC-type) | appr. 72 months
Quality of Life assessed by EORTC QLQ-C30. | appr. 72 months
Quality of Life assessed by EORTC QLQ-LC13. | appr. 72 months
Immune Effectors | appr. 72 months
  Changes in cellular and humoral immune effectors in peripheral blood and their correlation with response.
Mutational Landscape | appr. 72 months
  Mutational landscape of LCNEC in comparison to SCLC as well as squamous and Adenocarcinoma of the lung. The analysis will be using whole genome sequencing.
Tumor DNA (tDNA) level | appr. 72 months
  Dynamics of circulating tumor DNA levels (changes from baseline).
Therapy Resistance | appr. 72 months
  Mechanisms of therapy resistance (changes of immune invasion and mutational landscape in tumor re-biopsy upon progression).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wermke, Prof. Dr., Principal Investigator — Technische Universität Dresden (TUD)
Locations (15):
- Germany (15):
  - Charité - Universitätsklinikum Berlin Centrum 12, Medizinische Klinik, Berlin
  - Evangelische Lungenklinik, Berlin
  - Klinikum der Universität zu Köln, Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Dresden, Medizinische Klinik 1, Dresden
  - Klinikum der J.W. Goethe Universität, Medizinische Klinik II, Frankfurt am Main
  - Asklepios Fachkliniken München-Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Krankenhaus St. Elisabeth und St. Barbara Halle (Saale) GmbH, Halle
  - Thoraxklinik Heidelberg gGmbH, Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer des Deutschen Gemeinschafts-Diakonieverbandes GmbH, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum der Johannes Gutenberg Universität, III. Med. Klinik und Poliklinik, Mainz
  - Pius Hospital, Klinik für Hämatologie und Onkologie, Oldenburg
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - Rems-Murr-Klinikum Winnenden, Klinik für Hämatologie, Onkologie und Palliativmedizin, Winnenden